CLINICAL TRIAL: NCT00861198
Title: The Clinical Utility of Cholangioscopy and Pancreatoscopy in the Diagnosis and Management of Pancreaticobiliary Disorders
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: Pancreaticobiliary disorders
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Results first posted 2015-07-27 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-06

CONDITIONS: Disorders of the Pancreas and Biliary Tree
MeSH Terms: interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ERCP: Patients who have a medical indication for ERCP with cholangioscopy and/or pancreatoscopy and are referred for the procedure as part of their standard medical care will be considered for the study.
  Interventions: Other: ERCP as per medical indication

INTERVENTIONS:
Other: ERCP as per medical indication — ERCP as per medical indication

SUMMARY:
At the time of endoscopic retrograde cholangiopancreatography (ERCP) examination of the pancreaticobiliary system is done indirectly by radiologic means. Contrast is injected into the bile and/or pancreatic duct and outline of the duct is then viewed by fluoroscopic imaging. Frequently this is followed by diagnostic maneuvers (tissue acquisition) or therapeutic interventions (stone removal, stent insertion). Direct visualization of the bile and pancreatic ducts (cholangioscopy/pancreatoscopy) was developed 15 years ago and was shown to be superior to the indirect radiological view. The procedure did not become widely used secondary to high procedure related costs and equipment prone to failure. Recently a much improved (more affordable and more durable) cholangioscope was developed and approved by the FDA. The goal of this study is to prospectively record our experience with cholangioscopy and pancreatoscopy performed as medically indicated as part of standard medical care.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years or older.
* Scheduled to undergo ERCP with cholangioscopy and/or pancreatoscopy at the University of Florida, Gainesville, FL as medically indicated.
* Subject must be able to give informed consent

Exclusion Criteria:

* Any contraindication to ERCP.
* The subject is unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who have a medical indication for ERCP with cholangioscopy and/or pancreatoscopy and are referred for the procedure as part of their standard medical care will be considered for the study.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2006-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Draganov, MD, Principal Investigator — University of Florida, Division of Gastroenterology
Locations (1):
- Shands UF endoscopy Center, Gainesville, Florida, United States

REFERENCES:
- [Derived] Draganov PV, Lin T, Chauhan S, Wagh MS, Hou W, Forsmark CE. Prospective evaluation of the clinical utility of ERCP-guided cholangiopancreatoscopy with a new direct visualization system. Gastrointest Endosc. 2011 May;73(5):971-9. doi: 10.1016/j.gie.2011.01.003. Epub 2011 Mar 17. PMID 21419408

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 88 participants who were enrolled into the study; however, 13 were excluded because they did not qualify for the SpyGlass examination.
Groups:
- ERCP With Cholangioscopy and/or Pancretoscopy: Patients underwent ERCP and cholangiography or pancreatography with the Spyglass system.
Period: Overall Study
Arm/Group | ERCP With Cholangioscopy and/or Pancretoscopy
Started | 75
Completed | 70
Not Completed | 5
Not completed — SpyGlass Failed | 5

BASELINE CHARACTERISTICS:
Arm/Group | ERCP With Cholangioscopy and/or Pancretoscopy
Number analyzed (Participants) | 75
Age, Continuous [Mean (Full Range); unit: years] | 66 [22 to 96]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 38
Region of Enrollment [Number; unit: participants]
  United States | 75

OUTCOME MEASURES:

1. Primary Outcome: Successful Procedure Completion
Description: Defined based on the indication for SpyGlass. For cases involving biliary or pancreatic stones the procedure was considered successful when complete stone clearance was accomplished. For cases involving established or suspected nonstone-related lesions of the pancreatobiliary system, success was defined when all of the following criteria were met: successful advancement of the SpyScope to the desired target, adequate visualization of the area of interest and successful applications of all diagnostic and/or therapeutic maneuvers that were deemed necessary based on the endoscopic findings.
Time Frame: baseline
Measure: Number; unit: participants
Arm/Group | ERCP With Cholangioscopy and/or Pancretoscopy
Number analyzed (Participants) | 75
participants
  Successful completion | 70
  Unsuccessful/Failed | 5

ADVERSE EVENTS:
Time Frame: The reporting data was collected for 1 week after the procedure date
Arm/Group | ERCP
Serious Adverse Events (participants affected / at risk) | 0/75
Other Adverse Events (participants affected / at risk) | 0/75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes